CLINICAL TRIAL: NCT00865917
Title: Einfluss Selektiver I(f)-Blockade Auf Orthostase-Toleranz Und Sympathikusaktivität Bei Gesunden
Brief Title: Cardiovascular Effects of Selective I(f)-Channel Blockade
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Heidrum Mehling, Dr. med., Franz-Volhard-Centrum für Klinische Forschung
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CCB-CRC-07-02
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Adrenergic beta-Antagonists; Metoprolol; Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): beta-blocker
  Interventions: Drug: beta-blocker (Metoprolol)
- 2 (Experimental): I(f)-blocker
  Interventions: Drug: I(f)-blocker (ivabradine)
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: beta-blocker (Metoprolol) — Metoprolol 95 mg once per day
  Arms: 1
Drug: I(f)-blocker (ivabradine) — ivabradine 7.5 mg once per day
  Arms: 2
Drug: Placebo — matching appearance
  Arms: 3

SUMMARY:
The study compares three treatment modalities in a human model of Postural orthostatic tachycardia syndrome (POTS): beta-blockers, I(f)-blockers, and placebo.

DETAILED DESCRIPTION:
Elevated heart rate may lead to cardiac disease in the long-term. Therefore, drugs lowering heart rate are useful. Beta-blockers are an established treatment modality. They not only lower heart rate but also contractility, which might be undesirable in certain tachycardic disorders.

Postural orthostatic tachycardia syndrome (POTS) patients complain about dizziness, weakness, headache, lightheadedness, fatigue, nausea, and presyncope. In some patients there is elevated heart rate even during supine rest. In POTS patients it is preferable to lower heart rate without reducing cardiac contractility which can be achieved by using so-called I(f)-blockers. Thus, they might be superior to beta-blockers in POTS.

In our study, we artificially generate POTS in healthy male subjects for about 48 hours. We want to compare the cardiovascular effects and orthostatic tolerance of the following treatments: beta-blocker, I(f)-blocker, and placebo.

Moreover, we will quantify changes in cardiovascular autonomic regulation brought about by I(f)-blockade versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* age 18-40 years
* BMI: 18-30 kg/m²
* arterial blood pressure <=160/100 mm Hg
* co-operativity
* voluntariness

Exclusion Criteria:

* conditions in which treatment might be ineffective or insecure
* co-medication within the last 4 weeks
* participation in another clinical trial within the last 4 weeks
* unability to understand the study's aim
* drug or alcohol abuse
* secondary hypertension
* creatinine > 130 μM (1.47 mg/dl)
* GOT/GPT > 2 times normal
* GGT > 3 times normal
* contraindications against reboxetine, beta-blocker, ivabradine
* asthma, psoriasis
* diabetes
* heart failure (NYHA III or IV)
* coronary artery disease
* peripheral occlusive disease
* cerebrovascular disease
* ventricular extrasystoles (Lown III-V)
* atrial fibrillation
* resting heart rate <60/min
* neurologic/psychiatric disorder
* pulmonary hypertension
* dysthyroid metabolism

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Sub-study 'Orthostatic tolerance': Change in heart rate after 20 mins of passive orthostasis. Sub-study 'Sympathetic system': arterial pressure related heart rate | 12-18 hours

SECONDARY OUTCOMES:
'Orthostatic tolerance': Hemodynamics during head-up tilt. Time to presyncope. | 12-18 hours
'Sympathetic system': Muscle sympathetic nerve activity (MSNA). | 12-18 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Jordan, MD, Study Director — Hannover Medical School
Locations (2):
- Germany (2):
  - Franz-Volhard Centrum für Klinische Forschung, Berlin
  - Medizinische Hochschule Hannover, Hanover

REFERENCES:
- [Derived] Heusser K, Tank J, Brinkmann J, Schroeder C, May M, Grosshennig A, Wenzel D, Diedrich A, Sweep FC, Mehling H, Luft FC, Jordan J. Preserved Autonomic Cardiovascular Regulation With Cardiac Pacemaker Inhibition: A Crossover Trial Using High-Fidelity Cardiovascular Phenotyping. J Am Heart Assoc. 2016 Jan 13;5(1):e002674. doi: 10.1161/JAHA.115.002674. PMID 26764413
- [Derived] Zoerner AA, Schroeder C, Kayacelebi AA, Suchy MT, Gutzki FM, Stichtenoth DO, Tank J, Jordan J, Tsikas D. A validated, rapid UPLC-MS/MS method for simultaneous ivabradine, reboxetine, and metoprolol analysis in human plasma and its application to clinical trial samples. J Chromatogr B Analyt Technol Biomed Life Sci. 2013 May 15;927:105-11. doi: 10.1016/j.jchromb.2013.01.016. Epub 2013 Jan 29. PMID 23434314